CLINICAL TRIAL: NCT02765646
Title: eTryton Left Main Multi-center, Prospective, Non-randomized Single Arm Registry Evaluating the Tryton Side Branch Stent® for Treatment of de Novo CAD in Both LM and Circumflex (LCX) Coronary Arteries
Brief Title: eTryton Left Main Registry Tryton Side Branch Stent® Tmt of Denovo CAD in LM and CFX Arteries
Acronym: eTRYTONLM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tryton Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P0160
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Left Main Coronary Artery Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Coronary stent procedure (CSP)

SUMMARY:
The objective of this study is to demonstrate the clinical performance of the Tryton Side Branch Stent used in conjunction with a commercially available Drug Eluting Stent (DES) to treat de novo bifurcated lesions involving both the Left Main (LM) and Circumflex Coronary Artery(LCX).

DETAILED DESCRIPTION:
The registry study will involve the collection of demographic and clinical data, including in-hospital and follow-up data to determine primary composite endpoint of MACE (Major Adverse Cardiac Events) at 9 months and secondary endpoints. Secondary endpoints are defined as successful deployment of the Tryton stent and main vessel DES within the target lesion, angiographic success <30% residual stenosis in LM and LAD/LCX by visual estimate and TIMI 3 flow post procedure, and freedom of in-hospital MACE.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years old;
2. Patient is eligible for percutaneous coronary intervention (PCI);
3. Patient is an acceptable candidate for CABG;
4. Clinical evidence of ischemic heart disease and / or a positive functional registry. Documented stable angina pectoris (Canadian cardiovascular society classification (CCS) 1, 2, 3 or 4), unstable angina pectoris (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia;
5. Single high grade de novo bifurcation lesion with ≥50% and <100% stenosis in the distal part of left main, requiring stent placement across LCx Ostium, with TIMI flow > 2 by visual estimation;
6. The target lesion length must be able to be covered by a single main vessel stent ≥ 5.0mm and ≤ 32 mm in the main vessel and ≤ 32 mm in the side branch (visual estimate) and be covered by one Tryton stent and up to one DES in the side branch;
7. The reference vessel diameter of the main branch must be ≥ 2.5mm and ≤ 4.0 mm (visual estimate) and reference vessel diameter of the side branch must be ≥ 2.25mm and ≤ 3.5 mm (visual estimate);
8. If required by local regulations, the patient had been informed of the nature of the registry, agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee (MEC) of the respective clinical site;
9. The patient is willing to comply with follow-up evaluations.

Exclusion Criteria:

1. Female of childbearing potential;
2. Documented left ventricular ejection fraction (LVEF) ≤30%;
3. Evidence of an acute myocardial infarction within 48 hours of the intended treatment;
4. Known allergies to the following: Acetylsalicylic acid (ASA) (Aspirin®), Clopidogrel bisulfate (Plavix®.) or Ticlopidine (Ticlid®.), Heparin, contrast agent (that cannot be adequately pre-medicated);
5. Acute or chronic renal dysfunction (serum creatinine >2.0 mg/dl or >150μmol/L);
6. Target vessel has angiographic evidence of thrombus;
7. Previous interventional procedure (less than 1 year) anywhere within the left main artery including the bifurcation to the LAD and/or LCX;
8. Anticipated use of rotational atherectomy
9. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run offCONFIDENTIAL Page 7 of 18 August 11, 2015 - version 5 that will not be treated during the index procedure;
10. Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated;
11. Prior stent in the Left Main;
12. Prior stent within 5mm distal of the target lesion;
13. Total occluded dominant RCA;
14. Trifurcation lesion with a Ramus Intermedius diameter of >2.0 mm; a Diagonal Branch diameter of >2.0 mm within 5 mm of LAD origin; a Obtuse Marginal >2.0 mm diameter within 5 mm of LCx origin;
15. Patient is currently participating in an investigational drug or device registry that has not completed the primary endpoint or that clinically interferes with the current registry endpoints.
16. Stroke or transient ischemic attack within the prior 6 months;
17. In the Investigator's opinion patient has a co-morbid condition(s) that could limit the patient's ability to participate in the registry, compliance with follow-up requirements or impact the scientific integrity of the registry;
18. Recipient of heart transplant;
19. Life expectancy less than 1 year;
20. Braunwald Class IA, IIA and IIA angina pectoris;
21. Patients with severe congestive heart failure;
22. Patients with severe heart failure NYHA IV;-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CAD due to de novo stenotic lesion in the distal part of the LM at the bifurcation of the Left Anterior Descending Artery (LAD) and the Left Circumflex (LCX)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
MACE: cardiac death, non-index procedure related myocardial infarction, TLR, definite stent thrombosis | 9 months

SECONDARY OUTCOMES:
Procedural success: successful deployment of Tryton stent and MV DES within target lesion, Angiographic success <30% residual stenosis in LM and LAD/LCX bifurcation by visual est. and TIMI flow 3 post procedure and freedom of in-hospital MACE | 9 months
Clinical endpoints: MACE: total death, cardiac death, non-index procedure related MI, Target lesion revascularization (TLR), Target vessel revascularization (TVR), definite stent thrombosis, Procedure related MI | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Stylianos A Pyxaras, MD,FESC, Principal Investigator — Klinikum-Coburg, Germany
Locations (1):
- Klinikum Cobury GmbH, Coburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided